CLINICAL TRIAL: NCT06211257
Title: Phase 3 Superiority Trial Evaluating the Benefit of Dematerialized Information Media for Patients With Advanced Sarcomas Receiving Systemic Treatment for Metastatic or Locally Advanced Disease.
Brief Title: Superiority Trial Evaluating Digitalized Information Media for Patients With Advanced Sarcomas Receiving Systemic Treatment.
Acronym: ePPS-2202
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Canceropôle Nord Ouest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ePPS-2202; 2023-A00984-41 (Other: ANSM)
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Sarcoma Metastatic; Locally Advanced Soft Tissue Sarcoma
Keywords: Sarcoma; Advanced; Dematerialised; Care; Plan
MeSH Terms: conditions — Sarcoma; Neuroaxonal Dystrophies

STUDY DESIGN:
Intervention Model Description: Randomized 1:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group : standard PCP (No Intervention): Patient will receive standard support PCP
- Experimental group : demateralized PCP (Experimental): Patient will receive standard support PCP and dematerialized PCP (ePCP)
  Interventions: Other: Dematerialized Personalized Care Plan (ePCP)

INTERVENTIONS:
Other: Dematerialized Personalized Care Plan (ePCP) — Post-treatment support with standard support combined with dematerialized support
  Arms: Experimental group : demateralized PCP

SUMMARY:
ePPS-2202 is a study designed to evaluate the benefits of a dematerialised personalised care plan (PCP) compared to standard information/PCP for patients with advanced sarcomas receiving systemic treatment.

Participants will be randomised to an experimental group or a control group. Patients in the experimental group will receive the dematerialised PCP in addition to the standard PCP while patients in the control group will receive the standard PCP alone.

All patients will be followed until the end of second-line treatment, the start of a new line of treatment, or until the 24-month follow-up.

DETAILED DESCRIPTION:
ePPS-2202 is a phase 3, randomised,open-label, controlled, multicentre interventional study, designed to evaluate the benefits of a dematerialised personalised care plan (PCP) compared to standard information/PCP in patients with metastatic of locally advanced sarcomas with indication of a systemic treatment with pazopanib, tracbectedine, eribuline, ifosfamide or dacarbazine monotherapy.

Participants will be randomised to the experimental arm or the control arm. Patients in the experimental arm will receive the dematerialised PCP in addition to the standard PCP while patients in the control arm will receive the standard PCP alone.

All patients will be followed until the end of second-line treatment, the start of a new line of treatment, or until the 24-month follow-up.

The main analysis will compare the proportion of patients in each arm who experience at least one severe adverse event during the first 3 months of second-line treatment. Adverse events will be considered severe if they are graded 3 or higher according to NCI-CTCAE v5.0.

ELIGIBILITY:
Inclusion Criteria:

* Sarcomas of soft tissues or viscera ;
* Inoperable metastatic or locally advanced disease ;
* Indication for systemic treatment with pazopanib, trabectedine, eribulin, ifosfamide or dacarbazine monotherapy ;
* Patient covered by French social security ;
* Written, signed, informed consent ;

Exclusion Criteria:

* Prior inclusion in ePPS trial for a prior systemic treatment ;
* Poor understanding of French ;
* Difficulty accessing a computer ;
* Pregnant or nursing woman ;
* Person deprived of liberty or under guardianship ;
* Impossibility of undergoing medical follow-up for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Severe toxicity in the first 3 months of treatment | 3 months
  Severe toxicity will be assessed through the reporting of adverse events (AE). Will be considered as an AE all indesirable medical event regardless of the cause, occurring between randomisation and the end of treatment + 30days or the start of a new systemic anti-cancer treatment or the 24-month follow-up.
  All AE grade ≥ 3 according to Common Terminology Criteria for Adverse Events v5.0 scale (NCI-CTCAE) will be considered severe.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 24 months
  PFS will be defined as the time from randomisation to investigator-assessed disease progression (RECIST 1.1 or clinical). No progressive-patients will be censured at the 24-months follow-up.
Overall survival (OS) | 24 months
  OS will be defined as the time from randomisation to patient's death regardless of the cause. Alive patients will be censured at the 24-month follow-up.
Severe toxicity | 24 months
  Severe toxicity will be assessed through the reporting of adverse events (AE). Will be considered as an AE all indesirable medical event regardless of the relationship, occurring between randomization and the end of treatment + 30days or the stard of a new systemic anticancer treatment or the 24-month follow-up.
  All AE grade ≥ 3 according to Common Terminology Criteria for Adverse Events v5.0 scale (NCI-CTCAE) will be considered severe.
Nature of severe AEs | 24 months
  Description of the nature of severe adverse events occuring between randomization and the end of treatment + 30days or the start of a new systemic anticancer treatment or the 24-month follow-up, especially:
  * Asthenia ;
  * Gastrointestinal disorders: vomiting, anorexia, mucositis/aphthosis, diarrhea, constipation;
  * Skin disorders: hand-foot syndrome, phototoxicity, dry skin skin dryness;
  * Hypertension;
  * Hematological toxicity ;
  * Hematuric cystitis with ifosfamide;
  * Ifosfamide encephalopathy;
  * Extravasation with trabectedine;
AEs leading to hospitalization | 24 months
  Description of the adverse events leading to hospitalisation occuring between randomization and the end of treatment + 30days or the start of a new systemic anticancer treatment or the 24-month follow-up.
Survival weighted by quality of life | 24 months
  Survival weighted by quality of life with the "Quality adjusted Time Without Symptoms and Toxicit" method (Q-Twist)
Quality of life assessed by EORTC QLQ-C30 questionnaire | 3 months
  Quality of life assessed by "Quality of Life of Cancer Patients Questionnaire" (called EORTC QLQ-C30) at Baseline and at first oncological follow-up. The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.

CONTACTS AND LOCATIONS:
Overall Officials: Diane PANNIER, MD, Principal Investigator — Centre Oscar Lambret
Locations (11):
- France (11):
  - Centre Léon Bérard, Lyon, Auvergne-Rhône-Alpes
  - CHU Jean Minjoz, Besançon, Bourgogne-Franche-Comté
  - Centre Eugène Marquis, Rennes, Brittany Region
  - Centre Paul Strauss, Strasbourg, Grand Est
  - Centre Oscar Lambret, Lille, Hauts-de-France
  - CHU de Poitiers, Poitiers, Nouvelle-Aquitaine
  - Institut Claudius Regaud, Toulouse, Occitanie
  - Institut de Cancérologie de l'Ouest, Saint-Herblain, Pays de la Loire Region
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Hôpital Pitié-Salpêtrière AP-HP, Paris, Île-de-France Region
  - Gustave Roussy, Villejuif, Île-de-France Region